CLINICAL TRIAL: NCT00930150
Title: Cognitive Remediation in the Schizophrenia Trials Network
Brief Title: Feasibility of Providing Cognitive Remediation to People With Schizophrenia in a Clinical Network
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: T. Scott Stroup, MD, MPH, University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH090001-07; N01-MH090001-07; PCC: DSIR AT; N01MH090001 (NIH)
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posit Science Intervention (Experimental): Participants will receive targeted cognitive training and participate in a bridging group.
  Interventions: Behavioral: Targeted cognitive training; Behavioral: Bridging groups
- Control (Active Comparator): Participants will play commercially available computer games and participate in weekly groups to discuss health and wellness.
  Interventions: Behavioral: Computer control; Behavioral: Health and wellness groups

INTERVENTIONS:
Behavioral: Targeted cognitive training — Adaptive computer exercises that systematically increase in task difficulty as each participant's performance ability improves
  Arms: Posit Science Intervention
Behavioral: Computer control — Commercially available computer games selected based on quality, ability to hold interest, and lack of disturbing content
  Arms: Control
Behavioral: Bridging groups — Weekly group meetings that help participants apply their cognitive skills to everyday functioning, promote group identity, and promote socialization
  Arms: Posit Science Intervention
Behavioral: Health and wellness groups — Weekly group meetings that teach participants health and wellness skills
  Arms: Control

SUMMARY:
This study will test whether a cognitive remediation program to treat people with schizophrenia can be successfully implemented in a network of research clinics.

DETAILED DESCRIPTION:
Neurocognitive impairments, or problems with thinking and brain function, are a core component of schizophrenia. Such impairments, which can range from moderate to severe, are strongly associated with decreased benefit from psychiatric rehabilitation and problems with treatment adherence, socialization, employment, quality of life, and relapse. Researchers believe that the failure of medication to improve cognition may occur because medication treatment lacks cognitive stimulation. Cognitive remediation programs are a way to provide that stimulation, and they have shown moderate efficacy in improving cognition in people with schizophrenia. Implementing these cognitive remediation programs as part of schizophrenia treatment has occurred only at individual sites with highly trained research personnel. This study will test whether cognitive remediation programs for schizophrenia can be feasibly implemented at a network of sites that do not specialize in cognitive remediation research. This pilot study will gather preliminary efficacy data, but a larger study is required to draw definitive conclusions about treatment effects.

Participation in this study will last approximately 8 weeks. Participants will be randomly assigned to the Posit Science intervention group or the control group. Those in the Posit Science group will receive targeted cognitive training (TCT)-40 hours of adaptive computer exercises-and participate in a weekly bridging group that helps participants apply cognitive skills to everyday contexts. Length of the TCT may vary, depending on the availability of participants to complete the exercises. Those in the control group will play commercially available video games for the same number of hours and participate in a weekly health and wellness group. All participants will undergo assessments at baseline, mid-treatment, and post-treatment. Assessments will include self-report questionnaires and clinical interviews.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates adequate decisional capacity to make a choice about participating in the research study
* Diagnosis of schizophrenia or schizoaffective disorder, as defined by DSM-IV-TR criteria and confirmed by the Structured Clinical Interview for DSM-IV (SCID)
* Positive and Negative Syndrome Scale (PANSS) hallucinatory behavior, unusual thought content, and conceptual disorganization ratings of no greater than moderately severe (i.e., item scores must be less than or equal to 5)
* Meets all of the following cognitive performance and English language criteria:

  1. Learned English before age 12
  2. Able to complete the baseline Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) validly, based on the judgment of the investigator
  3. Raw score of 37 or greater on the Wide Range Achievement Test, reading subtest, 3rd edition (WRAT-3), used to establish minimum sixth grade reading level and estimated premorbid IQ
* Able to state specific goals relevant to the intervention that participant would like to achieve
* Able to participate in the computerized intervention, based on the judgment of the investigator

Exclusion Criteria:

* Psychiatric hospitalization within 8 weeks of random assignment
* Adjustment to antipsychotic treatment within 4 weeks of random assignment
* Currently taking an anticholinergic medication
* DSM-IV diagnosis of alcohol or substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months
* History of mental retardation, pervasive developmental disorder, or other neurological disorder (such as a traumatic brain injury, epilepsy, or Parkinson 's disease)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of a multisite trial using cognitive remediation | Measured at post-treatment

SECONDARY OUTCOMES:
Effect of cognitive remediation on functional outcomes, including change from baseline on UCSD Performance Based Skills Assessment (UPSA) total score, Specific Levels of Functioning (SLOF) total score, and Cognitive Assessment Interview (CAI) total score | Measured at post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Keefe, PhD, Principal Investigator — Duke University; T. Scott Stroup, MD, MPH, Principal Investigator — Columbia University
Locations (9):
- United States (9):
  - Yale University/Connecticut Mental Health Center, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Massachusetts, Worcester, Massachusetts
  - University of Minnesota School of Medicine, Minneapolis, Minnesota
  - The University of North Carolina, Chapel Hill, North Carolina
  - Philadelphia VA Medical Center-116A, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500
- [Derived] Keefe RS, Vinogradov S, Medalia A, Buckley PF, Caroff SN, D'Souza DC, Harvey PD, Graham KA, Hamer RM, Marder SM, Miller DD, Olson SJ, Patel JK, Velligan D, Walker TM, Haim AJ, Stroup TS. Feasibility and pilot efficacy results from the multisite Cognitive Remediation in the Schizophrenia Trials Network (CRSTN) randomized controlled trial. J Clin Psychiatry. 2012 Jul;73(7):1016-22. doi: 10.4088/JCP.11m07100. Epub 2012 May 15. PMID 22687548